CLINICAL TRIAL: NCT02725047
Title: The Effect of Cryotherapy in Pain Control, Function and Quality of Life in Individuals With Knee Osteoarthritis - Randomized Clinical Trial
Brief Title: The Effect of Cryotherapy in Pain Control, Function and Quality of Life in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Lucas Ogura Dantas, Lucas Ogura Dantas - Muscular Plasticity Laboratory - UFSCar, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRYO-123
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Cryotherapy; Thermotherapy; Hypothermia; Knee; Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Hyperthermia; Hypothermia | interventions — Cryotherapy; Ice; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TREATMENT - CRYOTHERAPY (Experimental): Patients with knee osteoarthritis, both sexes, with age between 40 and 75
  Interventions: Other: Cryotherapy
- PLACEBO - SAND (Placebo Comparator): Patients with knee osteoarthritis, both sexes, with age between 40 and 75
  Interventions: Other: Placebo - Sand

INTERVENTIONS:
Other: Cryotherapy — Crushed ice (1kg) inside a plastic bag (24x34x0,08 cm). The positioning of the plastic bags will cover the entire knee surface (Anterior, lateral and posterior region). After the positioning of the ice bags, they will be fixed with an elastic bandage (compression). To protect the skin against frost bites, all the knee surface will be covered with a moistened operative field (45x50x0,01 cm, 100% cotton)
  Other Names: Ice therapy
  Arms: TREATMENT - CRYOTHERAPY
Other: Placebo - Sand — Sand (1kg) inside a plastic bag (24x34x0,08 cm). The positioning of the plastic bags will cover the entire knee surface (Anterior, lateral and posterior region). After the positioning of the sand bags, they will be fixed with an elastic bandage (compression). Also, all the knee surface will be covered with a moistened operative field (45x50x0,01 cm, 100% cotton) to mimic the experimental group.
  Other Names: Placebo, sham
  Arms: PLACEBO - SAND

SUMMARY:
The purpose of this study is to verify the effect of cryotherapy in pain control, function and quality of life in individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
The purpose of this study is to verify the effect of cryotherapy in pain control, function and quality of life in individuals with knee osteoarthritis. This is a randomized controlled clinical trial, double-blinded. Will participate in the study 60 patients with knee osteoarthritis, diagnosed with clinical and radiographic criteria of the American College of Rheumatology, of both sexes, aged between 40 and 75 years. The total number of subjects will be divided randomly into two groups of 30 subjects each. During four consecutive days, for a period of 20 min, each group will receive one type of intervention around the knee with osteoarthritis: the cryotherapy group will receive an application of ice bags with compression and the placebo group will receive an application of sand bags with compression, the weight and volume of the sand bags will be similar to that used in cryotherapy. Every individual will have the following variables evaluated one day pre- and one day post-intervention: pressure pain threshold (Algometry), pain index (VAS), physical function questionnaires (WOMAC, KOOS) and physical activity (IPAQ). Two physical function tests will also be carried out: the 30s sitting and standing chair and the Timed Up and Go (TUG). Thermographic images will also be obtained for further temperature analysis of the knee with osteoarthritis. Moreover, after a period of 3 months, participants will perform a follow-up in which will be measured the VAS, WOMAC and KOOS questionnaires. Also, some Yes/No questions about the continued use of the therapy will be asked,

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis based on clinical and radiographic criteria of American College of Rheumatology
* Osteoarthritis signals in at least one of the compartments of the knee joint (tibiofemoral and / or the patellofemoral joint)
* Do not perform regular physical activity - less than three times a week regularly
* Grade 2 or 3 according to the criteria of Kellgren & Lawrence knee osteoarthritis radiographic examination scale.
* Minimum score of 4 cm in Visual Analogue Scale (total 10 cm)
* Body Mass Index less or equal to 45 kg/cm2

Exclusion Criteria:

* Physical therapy within 3 months prior to the research project
* Corticosteroid injection in the knee (in the previous 6 months)
* Medical condition (cardiorespiratory, neurological and / or musculoskeletal)
* Previous ankle, knee or hip surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (Pain scale): Change values from the pre evaluation to the post evaluation | The first measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  Visual Analog Scale for Pain:
  A visual analog scale (VAS) will be applied to measure the pain before and 1 day after the intervention. VAS is a well recognized tool to measure the intensity of pain that visually represents the intensity of pain that the individual believes to present. The scale will be positioned in front of the individual and will have a range of 0 to 10 cm, with 0 being the complete absence of pain and 10, the maximum intensity of pain reported by the individual.

SECONDARY OUTCOMES:
Thermography (Temperature device): Change values from the pre evaluation to the post evaluation | The second measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  A thermographic camera will be used (FLIR Systems Inc. model T-420) integrated with a real resolution of 320x240 pixels, sensors for measuring temperatures ranging from -20 °C (Celsius) to + 1200 °C and with a lower sensitivity to detect temperature differences of 0,08 ºC with ± 2°C of absolute temperature measurement, according to manufacturer's specifications (FLIR Systems Inc., 2006).
  The thermographic evaluation will be conducted in a controlled environment (21 °C ± 2 °C), with fluorescent lighting and a black background for the photos. Individuals will be advised not to bathe, perform physical exercise or use metabolic stimulants and decongestants 2 hours before the test, because these procedures affect the bloodstream and consequently the thermal images of interest. They will also be instructed not to use topical products like creams, powders or sprays on the area to be evaluated.
Algometry (Pressure pain threshold device): Change values from the pre evaluation to the post evaluation | The third measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  To measure the pressure pain threshold, it will be used a digital algometry of mechanical pressure (ITO Co., limited company (LTD)- Physiotherapy & Rehabilitation, OE-220 model, TOKYO, Japan) with a contact area of 1cm2. It will be performed 03 consecutive measurements (with an interval of 20s between each measurement) in 12 predetermined points chosen randomly. It will be used the average value of the 03 measurements (kg/s). At each point, the pressure pain threshold will be evaluated by applying the tip of a algometer at a speed of 1 kilogram per second, perpendicularly. The speed is controlled by the evaluator through the digital instrument display and the individual will receive a remote control with guidance to activate it at the exact moment that the pressure made by the algometry becomes painful. The interval time between each measurement will be observed to avoid temporal summation of cutaneous nociceptors.
WOMAC questionnaire (Self-administered questionnaire): Change values from the pre evaluation to the post evaluation | The fourth measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  All volunteers will answer to the questionnaire before and 1 day after the intervention. WOMAC is a self-report questionnaire designed to assess the problems experienced by people with OA of the lower limb. The score for the items is expressed through a Likert scale, where the rating is calculated as: none = 0, low = 25 = 50 moderate, severe = 75 and very severe = 100. The maximum score on each section is expressed as a percentage, with higher scores indicating greater pain, stiffness and physical dysfunction. Each point corresponds to a particular dimension (pain, stiffness and physical function). This questionnaire has been translated and validated for the Portuguese language from Brazil.
KOOS questionnaire (Self-administered questionnaire): Change values from the pre evaluation to the post evaluation | The fifth measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  All volunteers will answer to the questionnaire before and 1 day after the intervention. KOOS is a specific questionnaire which consists of 42 items divided into 5 subscales. It is self-administrative and aims to measure the quality of life and knee function evaluating five indicators: pain, other symptoms, function in daily life, function related to sports and recreation, and quality of life related to the knee. The answers are standardized (5 options for each question) and each question has a score ranging from 0 to 4. The initial score is transformed into a scale from 0 to 100, calculated for each subscale, so that higher values indicate better functionality and lower, a worse condition. It is also validated for the Portuguese language with acceptable psychometric characteristics when compared to the original one.
TUG (Timed up and go test:Physical function questionnaire): Change values from the pre evaluation to the post evaluation | The seventh measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  All volunteers will conduct the test before and 1 day after the intervention. TUG is a test that evaluates the balance of the individual in the sitting position, in sitting to standing transfers, stability in ambulation and gait course changes without the use of compensatory strategies. The test consists of asking the individual to stand from a chair, walk 3 meters, turn around, go back and sit back in the chair. The timing of the test is used as a functionally independent predictor: a time below 20 seconds is considered normal and above 30 seconds is considered as a possible increased risk of falls and functional dependency. It is estimated also the ability to get up, balance, posture, the base of gait (wide or short), the start of the march (if there is hesitation or freezing), speed, step size, continuity, symmetry, balance of the trunk and limbs, involuntary movements and the ability to return.
30 seconds chair stand test - : Physical function questionnaire: Change values from the pre evaluation to the post evaluation | The eighth measurement in the pre (First day - 1) and in the post (Last day - 6) evaluation - Full protocol - 6 days
  All volunteers performed the test before and 1 day after the intervention. The 30 seconds chair stand test is administered using an armless chair, with seat height of about 43cm from the ground. The chair has a rubber for not slipping under its support and is placed against a wall to avoid oscillations. The participant sits in the middle of the chair with the back straight, feet apart, aligned with the shoulder width apart and flat on the floor at an angle slightly behind the knee line. Moreover, to help maintain balance, one foot may be slightly placed ahead of the other and arms crossed against the chest. The test consists of the greatest number of times from a sitting position to a standing over a period of 30 seconds. Thus, it is possible to evaluate a wide range of skill levels with scores ranging from 0, for those who cannot complete a single repetition and values greater than 20 reps for the well prepared individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O Dantas, Ms. Student, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dantas LO, Breda CC, da Silva Serrao PRM, Aburquerque-Sendin F, Serafim Jorge AE, Cunha JE, Barbosa GM, Durigan JLQ, Salvini TF. Short-term cryotherapy did not substantially reduce pain and had unclear effects on physical function and quality of life in people with knee osteoarthritis: a randomised trial. J Physiother. 2019 Oct;65(4):215-221. doi: 10.1016/j.jphys.2019.08.004. Epub 2019 Sep 11. PMID 31521551